CLINICAL TRIAL: NCT06196268
Title: Effects of Core Strengthening and Pilates Exercises on Posture, Body Awareness, and Fatigue Among Female Athletes
Brief Title: Core Strengthening vs Pilates Exercises on Posture, Body Awareness and Fatigue Among Female Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR&AHS/23/0436
Record Dates: First submitted 2023-12-25; First posted 2024-01-09 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Exercise Movement Techniques; Muscle Strength; Athletes; Posture
Keywords: core strength; Pilates; Female Athletes; Posture; Fatigue
MeSH Terms: conditions — Fatigue | interventions — Exercise Movement Techniques

STUDY DESIGN:
Intervention Model Description: randomized clinical trail
Who Masked: Outcomes Assessor
Masking Description: the assessor who will take the readings is blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- core strengthening exercise (Experimental): Patients in Group A will receive core strengthening exercises along with the warm up exercises (lumbar stretches). CSE will constitute of abdominal hollowing, Side Bridge, supine extension bridge, straight leg rise from prone, alternate arm and leg raise from quadruped, and prone bridge. Total treatment will be of 60 mins with thrice a week for 6 weeks.
  Interventions: Other: core strengthening exercise
- Pilates exercise (Experimental): Patients in Group B will receive Pilates exercises along with warm up exercises which includes hundreds, one leg stretch, shoulder bridge, hip twist, scissors, side kicks. Total treatment will be of 60 mins with thrice a week for 6 weeks.
  Interventions: Other: Pilates exercise

INTERVENTIONS:
Other: core strengthening exercise — CSE will constitute of abdominal hollowing, Side Bridge, supine extension bridge, straight leg rise from prone, alternate arm and leg raise from quadruped, and prone bridge
  Arms: core strengthening exercise
Other: Pilates exercise — Pilates includes hundreds, one leg stretch, shoulder bridge, hip twist, scissors, side kicks
  Arms: Pilates exercise

SUMMARY:
The study is randomized and single-blinded. Ethical approval is taken from ethical committee of Riphah International University, Lahore. Participants who meet the inclusion criteria will be enrolled and allocated in group A & B through sealed envelope method by Non-probability Convenient random sampling technique. Subjects in Group A will receive Core Strengthening exercises. Group B will receive Pilates exercises.

DETAILED DESCRIPTION:
The objective of the study is to determine the Effects of Core Strengthening and Pilates Exercises on Posture, Body Awareness, and Fatigue among Female Athletes. The study is randomized and single-blinded. Ethical approval is taken from ethical committee of Riphah International University, Lahore. Participants who meet the inclusion criteria will be enrolled and allocated in group A & B through sealed envelope method by Non-probability Convenient random sampling technique. Subjects in Group A will receive Core Strengthening exercises. Group B will receive Pilates exercises. York posture rating chart, body awareness scale, and modified fatigue impact scale will be done at the baseline and after the completion of treatment at 6 weeks.

The data will be analyzed by SPSS, version 25. Statistical significance is P=0.05.

ELIGIBILITY:
Inclusion Criteria:

* Amateur female athletes 18-26 years of age,
* Duration of playing at least 6 months to 1 year,
* BMI <29 kg/m2, Core training not less than 4 weeks,
* Females having no previous injury that could interfere with the study,
* Females are not currently using nutritional supplements

Exclusion Criteria:

* Smoking,
* sleeping medications,
* complementary medicine use over the last six months,
* Stressful events in the past three months,
* presence of a physical or mental illness, or surgical history,
* Presence of any neurological and vascular disease,
* Participants having another exercise program which can affect the results,
* Participants who are not able to participate in any regular exercise program.

Ages: 18 Years to 26 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — participant should be healthy female
Enrollment: 44 (Actual)
Dates: Start 2023-10-20 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2024-02-20 (Actual)

PRIMARY OUTCOMES:
Posture | pre and 6 weeks post interventional
  posture of the female athlete will be measured by New York posture rating chart for each of 13 body alignment segments
Body Awareness | pre and 6 weeks post interventional
  Body Awareness Questionnaire will be used to measure the body awareness of female athlete
Fatigue | pre and 6 weeks post interventional
  Modified fatigue impact scale instrument provides an assessment of the effects of fatigue with scoring from 36 in 21 items

CONTACTS AND LOCATIONS:
Overall Officials: Eiza Shamshad, DPT, Principal Investigator — Study Principal Investigator
Locations (1):
- Pakistan sports board, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gandolfi M, Vale N, Dimitrova E, Zanolin ME, Mattiuz N, Battistuzzi E, Beccari M, Geroin C, Picelli A, Waldner A, Smania N. Robot-Assisted Stair Climbing Training on Postural Control and Sensory Integration Processes in Chronic Post-stroke Patients: A Randomized Controlled Clinical Trial. Front Neurosci. 2019 Oct 24;13:1143. doi: 10.3389/fnins.2019.01143. eCollection 2019. PMID 31708735
- [Background] Martins HS, Ludtke DD, Cesar de Oliveira Araujo J, Cidral-Filho FJ, Inoue Salgado AS, Viseux F, Martins DF. Effects of core strengthening on balance in university judo athletes. J Bodyw Mov Ther. 2019 Oct;23(4):758-765. doi: 10.1016/j.jbmt.2019.05.009. Epub 2019 May 14. PMID 31733759
- [Background] Gungor F, Tarakci E, Ozdemir-Acar Z, Soysal A. The effects of supervised versus home Pilates-based core stability training on lower extremity muscle strength and postural sway in people with multiple sclerosis. Mult Scler. 2022 Feb;28(2):269-279. doi: 10.1177/13524585211012202. Epub 2021 Apr 28. PMID 33908294
- [Background] de Jong M, Lazar SW, Hug K, Mehling WE, Holzel BK, Sack AT, Peeters F, Ashih H, Mischoulon D, Gard T. Effects of Mindfulness-Based Cognitive Therapy on Body Awareness in Patients with Chronic Pain and Comorbid Depression. Front Psychol. 2016 Jun 30;7:967. doi: 10.3389/fpsyg.2016.00967. eCollection 2016. PMID 27445929
- [Background] Goldberg SB, Tucker RP, Greene PA, Davidson RJ, Wampold BE, Kearney DJ, Simpson TL. Mindfulness-based interventions for psychiatric disorders: A systematic review and meta-analysis. Clin Psychol Rev. 2018 Feb;59:52-60. doi: 10.1016/j.cpr.2017.10.011. Epub 2017 Nov 8. PMID 29126747
- [Background] Clark DR, Lambert MI, Hunter AM. Contemporary perspectives of core stability training for dynamic athletic performance: a survey of athletes, coaches, sports science and sports medicine practitioners. Sports Med Open. 2018 Jul 16;4(1):32. doi: 10.1186/s40798-018-0150-3. PMID 30014195
- [Background] Mitchell UH, Johnson AW, Adamson B. Relationship between functional movement screen scores, core strength, posture, and body mass index in school children in Moldova. J Strength Cond Res. 2015 May;29(5):1172-9. doi: 10.1519/JSC.0000000000000722. PMID 25719919
- [Background] Karuc J, Misigoj-Durakovic M. Relation between Weight Status, Physical activity, Maturation, and Functional Movement in Adolescence: An Overview. J Funct Morphol Kinesiol. 2019 May 30;4(2):31. doi: 10.3390/jfmk4020031. PMID 33467346